CLINICAL TRIAL: NCT05983237
Title: Phase Ib Study of Fluzoparib in Combination With Camrelizumab and Temozolomide in Advanced Melanoma With Homologous Recombination (HR) Mutation ，a Single-center Open-label Exploratory Clinical Trial
Brief Title: Fluzoparib in Combination With Camrelizumab and Temozolomide in Advanced Melanoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jun Guo (Other)
Responsible Party: Sponsor-Investigator, Jun Guo, Director, Peking University Cancer Hospital & Institute
Organization: Peking University Cancer Hospital & Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-MM-Ⅱ-005
Record Dates: First submitted 2023-07-11; First posted 2023-08-09 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Melanoma
Keywords: Homologous recombination (HR); PARP inhibitor; anti PD-1 antibody
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camre+Fluzo+TMZ (Experimental): This arm will enroll patients who has advanced melanoma with a genetic HR mutation/ alteration .
  Interventions: Drug: Fluzoparib Camrelizumab Temozolomide

INTERVENTIONS:
Drug: Fluzoparib Camrelizumab Temozolomide — Fluzoparib 50-150mg bid po, d1-21, q3w Camrelizumab 200mg iv, d1, q3w Temozolomide 50mg/m2-200mg/m2 d1-5,q3w

SUMMARY:
The purpose of this study is to evaluate how well fuzoparib in combination with camrelizumab and temozolomide works in treating patients with advanced, metastatic melanoma with the homologous recombination (HR) pathway gene mutation / alteration.

DETAILED DESCRIPTION:
Treatment with PARP inhibitors could represent a novel opportunity to selectively kill a subset of cancer cells with deficiencies in DNA repair pathways. Non-BRCA deficiencies in homologous recombination DNA repair genes could also enhance tumor cell sensitivity to PARP inhibitors. Therefore, PARP inhibitors are also selectively cytotoxic for cancer cells with deficiencies in DNA repair proteins other than BRCA1 and BRCA2.

In melanoma, genetic HR mutation/ alterations are rather common. Retrospective data showed that nearly18-40% of melanoma harbors a mutation in at least 1 of the HR genes in their tumor. The commonly altered genes were ARID1A, FANCA, ATM, BRCA1, ATRX and BRCA2, ATR, BRCA1 BRIP1 and SF3B1. These findings indicate that HR mutations / alterations are frequently observed in metastatic melanoma, and they suggest that PARP inhibitors could potentially be of a great clinical value in a substantial portion of the patients with advanced melanoma.

In this clinical study, clinical efficacy of fluzoparib in combination with camrelizumab and temozolomide will be evaluated by assessing an objective clinical response rate in patients with advanced, metastatic melanoma with the homologous recombination (HR) pathway gene mutation / alteration.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of unresectable or metastatic stage III or IV melanoma;
2. Must have genetic HR and/or SF3B1 mutation/ alteration;
3. Must have measurable disease based on RECIST 1.1;
4. Must have an ECOG performance status of 0 to 1;
5. Must have recovered from all AEs due to previous therapies to ≤Grade 1 or baseline;
6. Anticipated overall survival more than 3 months;
7. Male and no pregnant female, able to adapt birth control methods during treatment.

Exclusion Criteria:

1. Previously treated with a PARP inhibitor;
2. Hypersensitivity to Fluzoparib or Camrelizumab or Temozolomide;
3. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug;
4. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug;
5. Patients with a history of other (including unknown primary) malignancies within 5 years prior to the first dose of trial treatment;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-08-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 6 months
  ORR of Fluzoparib in combination with Camrelizumab and Temozolomide in patients with advanced melanoma with genetic homologous recombination (HR) mutation/ alteration using RECIST v1.1

CONTACTS AND LOCATIONS:
Overall Officials: Jun Guo, Study Director — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, China